CLINICAL TRIAL: NCT01507870
Title: Randomized Controlled Prospective Multicenter Study Primary Onlay- Mesh After Elective Median Laparotomy in Patients With BMI ≥ 27
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Austrian Hernia Study Group (Other)
Responsible Party: Principal Investigator, PD Dr. Herwig Pokorny, Principal Investigator, Austrian Hernia Study Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Primary Onlay
Record Dates: First submitted 2012-01-05; First posted 2012-01-11 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-07

CONDITIONS: Incisional Hernia; Obesity
Keywords: body mass index
MeSH Terms: conditions — Incisional Hernia; Obesity

ARMS (2):
- prophylactic onlay mesh (Active Comparator)
  Interventions: Procedure: onlay mesh placement
- continuous running suture (No Intervention): continuous running suture of the linea alba

INTERVENTIONS:
Procedure: onlay mesh placement — prophylactic onlay mesh in patients with median laparotomy
  Arms: prophylactic onlay mesh

SUMMARY:
Incisional hernia is one ot the most frequently seen long term complications in abdominal surgery. Despite studies on the optimal suturing technique for laparotomies, the risk for incisional hernia after midline incision remains about 5-20 %. One major risk factor for incisional hernia after a median laparotomy is obesity.

The closure technique of midline incisions has remained unchanged since many decades and primarily consists of suturing the linea alba. Interest in prevention of incisional hernias with the aid of synthetic mesh is growing and only one large randomized trial is active recruiting patients in Germany, Netherlands and Belgium (Prima Trial).

Patients with a BMI of more than 27 have a high risk of developing an incisional hernia after midline incision with an incidence of 22% after 12 months. This high risk group of patients may benefit from prevention.

Some small studies have been performed to evaluate the usefulness and safety of primary laparotomy wound closure with the aid of prosthetic mesh. These studies show a very low risk for incisional hernias and a low infection rate, even when used in contaminated wounds such as colostomy surgery.

The goal of this study is to evaluate the effectiveness of incisional hernia prevention after elective median laparotomy in patients with a BMI of more than 27. A randomized controlled trial will be performed comparing the commonly used technique of running suture to close with the aid of a prosthetic onlay mesh. The primary outcome measure will be incisional hernia occurrence. Secondary outcome measures will be complications, surgical site infections, post-operative pain and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Every elective midline laparotomy for patients with a BMI of more than 27. Signed informed consent

Exclusion Criteria:

* Age < 18 years
* Emergency procedure
* Inclusion in other trials
* Previous midline incision
* Life expectancy less than 24 months
* Pregnant women
* Immune suppression therapy within 2 weeks before surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
incisional hernia occurrence | 3 years

SECONDARY OUTCOMES:
complications | 3 years
  haematoma formation, seroma formation, surgical site infection (SSI - classification)
postoperative pain | 14 days postoperative
  VAS
life quality | 14 days postoperative
  MOS SF-36

CONTACTS AND LOCATIONS:
Locations (1):
- Wiener Neustadt, Lower Austria, Austria